CLINICAL TRIAL: NCT05265351
Title: Ultrafast Ultrasound for the Functional Assessment of the Diaphragm: Agreement With Standards Mechanical and Electrophysiological Variables and Diagnosis Performance
Brief Title: Ultrafast Ultrasound for the Functional Assessment of the Diaphragm
Acronym: ECHOSTIM-EFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHOSTIM-EFR
Record Dates: First submitted 2022-02-01; First posted 2022-03-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diaphragm Dysfunction
Keywords: Diaphragm; Ultrafast ultrasound imaging; Electrophysiology; Cervical magnetic stimulation; Electromyography

STUDY DESIGN:
Intervention Model Description: Patients with confirmed or suspected diaphragm dysfunction undergoing transdiaphragmatic pressure measurement in response to phrenic neurostimulation as part of their follow-up or diagnostic. During this examination, ultrafast ultrasound imaging will be performed in diaphragm to capture elicited responses to assess the relationship between the variables derived from the ultrasound of the diaphragm and the variables usually measured during the evaluation of the transdiaphragmatic twitch pressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with confirmed or suspected diaphragm dysfunction (Experimental): Diaphragm function will be assess. Surface electromyography of the diaphragm will be performed in parallel. The abdominals displacement will be recorded using strain gauge. The intra-thoracic and intra-abdominal pressure will be measured using esophageal and gastric catheter-balloon.
  Ultrafast ultrasound imaging will be performed during Cervical and bi-lateral anterior magnetic stimulation, and during phrenic electrical stimulation.
  Interventions: Diagnostic Test: Transdiaphragmatic pressure measurement; Diagnostic Test: EMG

INTERVENTIONS:
Diagnostic Test: Transdiaphragmatic pressure measurement — Ultrafast ultrasound imaging of the diaphragm during artificially evoked responses
  Other Names: Ultrafast ultrasound imaging
Diagnostic Test: EMG — Surface electromyography of the diaphragm for phrenic nerve conduction study

SUMMARY:
The aims of the current study are as follows:

i) Investigate the relationships between indices derived from ultrafast ultrasound imaging and Pditw, ii) Investigate the relationships between indices derived from ultrafast ultrasound imaging and diaphragm EMG, iii) Investigate the performance of ultrafast ultrasound for the diagnosis of diaphragm dysfunction, iv) Investigate the ability of ultrafast ultrasound imaging to decipher the cause of diaphragm dysfunction i.e. contractility alteration and/or phrenic nerves conduction defect.

DETAILED DESCRIPTION:
The Neuromuscular Physiology and Evaluation Laboratory of the Institute of Myology recently reported that artificially stimulated diaphragm contraction may be captured and quantified using ultrafast ultrasound imaging. By filming the diaphragm at very high frame rate, one may extract ultrasound indices such as diaphragm thickening fraction and diaphragm tissue velocity. The same team showed that these indices, in particular, maximal diaphragm tissue velocity were strongly reliable and related to Pditw in healthy subjects. This approach bridges the gap between non-volitional (that are commonly combined with internal pressure measurements) and non-invasive procedures. Whether the relationships between indices derived from ultrafast ultrasound and Pditw exist in patients presenting with actual or suspicion of diaphragm dysfunction remains to be specifically investigated. Similarly, the potential of this approach for the diagnosis of phrenic conduction abnormalities remains to be assessed as it may help to circumvent confounding factors associated with surface EMG.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Patients with confirmed diaphragm dysfunction or suspicion
* Written informed consent
* Able to comply with all protocol requirements
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Known allergy to latex
* Known allergy to Lidocaine or similar product
* Pacemaker
* Guardianship/trusteeship
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Significant relationship between maximal diaphragm tissue velocity and transdiaphragmatic twitch pressure | Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Significant relationship between the diaphragm tissue latency and EMG latency | Through study completion, an average of 6 months
Accurate discrimination between patients with or without diaphragm dysfunction using metrics derived from ultrafast ultrasound | Through study completion, an average of 6 months
Accurate discrimination between patients with or without phrenic conduction abnormality using metrics derived from ultrafast ultrasound | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Damien BACHASSON, PhD, Principal Investigator — Institute ofMyology
Locations (1):
- Département R3S - Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No